CLINICAL TRIAL: NCT03055130
Title: HPV Infection and Cervical Neoplasm in Women With Inflammatory Bowel Disease: a Cross-sectional Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiang Gao, Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: HHBY-YJFA-20160813
Record Dates: First submitted 2017-02-08; First posted 2017-02-16 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: HPV-Related Cervical Carcinoma; Inflammatory Bowel Diseases; Cervical Neoplasm
MeSH Terms: conditions — Inflammatory Bowel Diseases; Uterine Cervical Neoplasms | interventions — Thrombin Time

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week

GROUPS / COHORTS (2):
- Case group: Female IBD patients who had sexual life between 21-60 years-old were recruited.
  Interventions: Other: Thinprep Cytology Test (TCT) and HPV infection types were tested by gynecologist
- control group: Female people who perform physical examination in our hospital between 21-60 years-old were recruited as control during the study period.
  Interventions: Other: Thinprep Cytology Test (TCT) and HPV infection types were tested by gynecologist

INTERVENTIONS:
Other: Thinprep Cytology Test (TCT) and HPV infection types were tested by gynecologist

SUMMARY:
The associations between female inflammatory bowel disease (IBD) patients and human papilloma virus (HPV) infection and cervical neoplasia (dysplasia or cancer) were unclear. Especially there was no data for Chinese IBD population. So we investigated the incidence and risk factors of HPV infection and cervical neoplasia (dysplasia or cancer) in female IBD patient.

ELIGIBILITY:
Inclusion Criteria:

1. between 20-60 years old;
2. Patients diagnosed as IBD according to previously established international criteria

Exclusion Criteria:

1. Patients refuse to participating

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All consecutive female adult patients betwween 20-60 year old were recruited from July 2015 to July 2017. Female persons who performed physical examination in our hospital with the same age were recuited as control. All of the received HPV DNA testing and TCT. The case and control were matched 1:3
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2017-05 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
The different infection rate of HPV between controls and patients by detecting HPV-DNA using reverse dot-blot method. | July 2015 to July 2017
  The difference of infection rate of HPV between healthy control and IBD patients was not clear.We are detecting HPV-DNA by reverse dot-blot and calculate the positive rate of HPV infection among controls and patients.
The different incidence of cervical neoplasm between controls and patients by performing Thinprep Cytology Test | July 2015 to July 2017
  The difference of the incidence of cervical neoplasm between healthy control and IBD patients was not clear.All the controls and patients are going to perform Thinprep Cytology Test which could detect intraepithelial neoplasia of cervix.

SECONDARY OUTCOMES:
Find drugs relating to HPV infection of IBD patients | July 2015 to July 2017
  Most IBD patients used steroid, infliximab or immunosuppressant to manage the disease. We separate patients into two groups according to using a certain drug or not. Then we compare the HPV infection rate between the two groups by Pearson-X2 test using SPSS 13.0 software (SPSS Inc., Chicago, Ill., USA).P < 0.05 was considered statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Gao, PhD, Study Director — The sixth affiated hospital of Sun-Yat sen University
Locations (1):
- Department of Gastroenterology, Guangzhou, Guangdong, China